CLINICAL TRIAL: NCT03756402
Title: The Relationship Between IRRIV and RFR Under Normal Conditions: External Validation
Brief Title: External Validation of IRRIV Test Relationship With Renal Functional Reserve
Acronym: IRRIV-RFR
Status: Completed | Type: Observational
Sponsor: Ospedale San Bortolo di Vicenza (Other)
Responsible Party: Principal Investigator, Sara Samoni, Medical Doctor, Ospedale San Bortolo di Vicenza
Other Study IDs: 0103/15
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; ColorDoppler; IRRIV test; Renal functional reserve; Renal resistive index; Ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Subjects: All subjects underwent protein loading test and IRRIV test on the same day. The renal resistive index (RRI) measurements were performed by one trained sonographer using a multi-frequency convex probe through a manual RRI calculations. The RRIs were measured on three interlobular arteries (superior, middle and inferior) in each kidney, and expressed as a mean value. RFR was measured using an oral protein loading test and was then defined as the difference between the highest CrCl obtained after the protein load and the baseline CrCl measured on rest conditions. Urinary creatinine and sCr were measured by the enzymatic method (IL testTM Instrumentation(R), Laboratory SpA, Milano, Italy) and by ILab650 (Instrumentation Laboratory, Werfen Group, Barcelona, Spain).

SUMMARY:
The assessment of renal functional reserve (RFR) has been proposed for the risk stratification of patients undergoing potentially nephrotoxic procedures. The investigators hypothesized that there is a correlation between IRRIV and RFR under normal conditions. For this purpose, externally validation of IRRIV test is performed in a validation cohort of healthy subjects.

DETAILED DESCRIPTION:
Normal subjects display a significant capacity to increase in baseline GFR under physiological needs (e.g. pregnancy) or pathological states (e.g. solitary kidney). This capacity is known as renal functional reserve (RFR), and it is calculated as the difference between the measured maximum GFR achieved through a renal stress test and the baseline GFR measured in rest conditions.In clinical practice, the most common renal stress test is performed as a standardized protein loading test. In a pilot study, the investigators demonstrated a significant correlation between RFR and the intra-parenchymal renal resistive index variation (IRRIV) during an echo renal stress test in a cohort of healthy volunteers. IRRIV test has proven to be rapid, safe, bedside and easy to perform and it might represent a preliminary test in screening patients' RFR. For this purpose, externally validation of IRRIV test is performed in a validation cohort of healthy subjects.

ELIGIBILITY:
Inclusion criteria were:

* Age more than 18 years old;
* Baseline estimated GFR, calculated using the chronic kidney disease epidemiology collaboration (CKD-EPI) equation, greater than or equal to 60 ml/min/1.73 m2.

Exclusion criteria were:

* Age less than 18 years old;
* Comorbidities potentially affecting renal function (i.e. arterial hypertension, diabetes, vasculopathy, etc.;
* Chronic administration of drugs able to modify renal blood flow and/or GFR (angiotensin converting enzyme-inhibitors (ACEI), angiotensin receptor blockers (ARB), calcium channel blockers, loop diuretics etc.);
* Pregnancy;
* Ultrasound evidence of morphological kidney abnormalities and/or renal artery stenosis;
* Nonsteroidal anti-inflammatory drugs (NSAIDs) or contrast media in the 2 days before the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects undergoing a protein loading and IRRIV test evaluation
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-01-10 (Actual)

PRIMARY OUTCOMES:
Externally validate IRRIV test | Change from baseline to 60 minutes
  A weight of 10% of the patient's body weight was applied on the abdomen. RRIs were recorded in a middle interlobular artery, every minute for 10 minutes during the echo-renal stress test. The lowest RRI reached was taken as reference (stress RRI). The IRRIV was defined as the percentage difference between baseline RRI and stress RRI.

SECONDARY OUTCOMES:
Correlation between IRRIV test and RFR | Change from baseline to 60 minutes
  Correlation between IRRIV and RFR is tested through a Pearson analysis. Concordance between presence of RFR (i.e. a RFR≥15ml/min/1.73m2) and a positive/uncertain/negative IRRIV is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, MD, Study Director — Ospedale San Bortolo di Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Samoni S, Nalesso F, Meola M, Villa G, De Cal M, De Rosa S, Petrucci I, Brendolan A, Rosner MH, Ronco C. Intra-Parenchymal Renal Resistive Index Variation (IRRIV) Describes Renal Functional Reserve (RFR): Pilot Study in Healthy Volunteers. Front Physiol. 2016 Jul 6;7:286. doi: 10.3389/fphys.2016.00286. eCollection 2016. PMID 27458386
- See also: PPT SSamomi — https://www.youtube.com/watch?v=9V4RoWvL9cs